CLINICAL TRIAL: NCT04433611
Title: Analgesic Efficacy of Intrauterine Lidocaine Flushing in Hysterosalpingo-foam Sonography: A Double-blind Randomized Controlled Trial
Brief Title: Efficacy of Uterine Lidocaine Flushing in HyFoSy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: # 0189-19
Record Dates: First submitted 2020-06-07; First posted 2020-06-16 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-05

CONDITIONS: To Evaluate the Efficacy of Flushing the Uterine Cavity With Lidocaine Before Hysterosalpingo-Foam Sonography to Reduce Procedure-related Pain
MeSH Terms: interventions — Lidocaine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 'lidocaine flushing' group (Experimental): intrauterine infusion of 2% lidocaine (Rafa laboratories, Israel) just prior to HyFoSy
  Interventions: Drug: 2% lidocaine
- Placebo group (Placebo Comparator): intrauterine infusion of 0.9 % normal saline (placebo group) just prior to HyFoSy.
  Interventions: Drug: 0.9 % normal saline

INTERVENTIONS:
Drug: 2% lidocaine — intrauterine infusion of 2% lidocaine (Rafa laboratories, Israel) just prior to HyFoSy
  The VAS consisted of a 10 cm line ranging from 0 to 10 (anchored by 0=no pain and 10=very severe pain). Patients were asked to mark the number that represented their perceived level of pain. Based on the VAS scores, the pain level ratings were classified as: mild (rated 1-3), moderate (4-6) or severe (7-10).
  Arms: 'lidocaine flushing' group
Drug: 0.9 % normal saline — intrauterine infusion of 0.9 % normal saline
  Arms: Placebo group

SUMMARY:
To evaluate the efficacy of flushing the uterine cavity with lidocaine before Hysterosalpingo-Foam Sonography (HyFoSy) to reduce procedure-related pain.

DETAILED DESCRIPTION:
This randomized, double-blind, placebo-controlled trial was approved by the institutional ethics committee (# 0189-19; approval 22-09-2019) and written informed consent was obtained from all participants. The sample was composed of women who were referred for tubal patency evaluation as part of their fertility workup. Exclusion criteria were a known allergy to lidocaine, unprotected intercourse, profuse vaginal bleeding and genital tract inflammation or infections (e.g. pelvic inflammatory disease (PID) or suspected sexually transmitted diseases (purulent vaginal discharge upon speculum insertion), salpingitis or tubo-ovarian abscess), psychological or neurological lesions affecting sensation, prior cervical surgery, cervical stenosis.

Randomization took place on the day of the procedure so that the staff had sufficient time to prepare the instruments and the medication/placebo. Women were randomized into one of two groups in a 1:1 ratio, using a predetermined randomization code, prepared by a research nurse. They were allocated to receive either: (1) an intrauterine infusion of 2% lidocaine (Rafa laboratories, Israel) ('lidocaine flushing' group), or (2) an intrauterine infusion of 0.9 % normal saline (placebo group) just prior to HyFoSy.

An assigned nurse prepared the medications according to the allocation group. Lidocaine and normal saline were placed in identical 10-mL disposable syringes. The lidocaine solution as well as the normal saline were both colorless and thus indistinguishable by the women and the performing sonographer, all of whom were blind to the group assignment.

No form of premedication was given before HyFoSy. The exam was performed after complete cessation of menstrual bleeding and before the 14th day of the ovulatory cycle. The women were placed in the supine position on an examination couch and a baseline transvaginal scan was performed by one of two experienced clinicians to detect any pelvic pathologies. A vaginal speculum was introduced into the vagina for visualization of the cervix. The cervix and vagina were cleansed with iodine solution. A balloon-less GIS catheter (GynaecologIQ)19 with a soft tapered tip was inserted into the endocervical canal for all HyFoSy procedures. The use of a tenaculum for uterine traction or a cervical dilatator to introduce the catheter was avoided in all cases. The speculum was then removed, taking care not to dislodge the catheter, and the ultrasound transducer was introduced vaginally. The abovementioned phase of the exam was performed by the same physician in all cases. The un-labelled solution (2% lidocaine solution or normal saline) was instilled slowly into the uterine cavity through the catheter until good distension and clear visualization of the uterine cavity was obtained. The ExEm® Foam-kit was used to produce foam according to the manufacturer's instructions9. The foam was then injected slowly via the GIS catheter under direct ultrasound guidance, until its passage or non-passage through both fallopian tubes had been assessed. All examinations were performed using a Samsung WS80A ultrasound system equipped with a V5-9 MHz endovaginal probe.

Pain scores were obtained before the procedure to collect a baseline value and were reassessed after the HyFoSy examination. All patients were asked to stay for 10-20 min in a waiting area and were asked to score the level of pain they experienced during the procedure on a visual analog scale (VAS) as described in20. The VAS consisted of a 10 cm line ranging from 0 to 10 (anchored by 0=no pain and 10=very severe pain). Patients were asked to mark the number that represented their perceived level of pain. Based on the VAS scores, the pain level ratings were classified as: mild (rated 1-3), moderate (4-6) or severe (7-10).

Sample size was calculated to detect 1 unit of mean difference of pain score between the two groups using the VAS, assuming that 1 was the SD (standard deviation) within the group. Twenty-seven women were needed in each group to reject the null hypothesis of 0.05 with a power of 0.9. Adding 30% to that number to compensate for any missing data gave a number of 39 women in each group.

ELIGIBILITY:
Inclusion Criteria:

*all women who were referred for tubal patency evaluation as part of their fertility workup.

Exclusion Criteria:

* known allergy to lidocaine.
* unprotected intercourse.
* profuse vaginal bleeding and genital tract inflammation or infections (e.g. pelvic inflammatory disease (PID).
* suspected sexually transmitted diseases (purulent vaginal discharge upon speculum insertion), salpingitis or tubo-ovarian abscess).
* psychological or neurological lesions affecting sensation, prior cervical surgery, cervical stenosis.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2020-06-17 (Actual); Primary Completion 2020-10-01 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
visual analog scale (VAS) pain score | 22 months
  The VAS consisted of a 10 cm line ranging from 0 to 10 (anchored by 0=no pain and 10=very severe pain). Patients were asked to mark the number that represented their perceived level of pain. Based on the VAS scores, the pain level ratings were classified as: mild (rated 1-3), moderate (4-6) or severe (7-10).

CONTACTS AND LOCATIONS:
Overall Officials: Yaakov Melcer, Principal Investigator — Assaf-Harofeh Medical Center
Locations (1):
- Yaakov Melcer, Yavné, Select A State Or Province, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Analytic Code
Time Frame: 1 year

REFERENCES:
- [Derived] Melcer Y, Nimrodi M, Levinsohn-Tavor O, Gal-Kochav M, Pekar-Zlotin M, Maymon R. Analgesic Efficacy of Intrauterine Lidocaine Flushing in Hysterosalpingo-foam Sonography: A Double-blind Randomized Controlled Trial. J Minim Invasive Gynecol. 2021 Aug;28(8):1484-1489. doi: 10.1016/j.jmig.2020.11.019. Epub 2020 Nov 26. PMID 33249268